CLINICAL TRIAL: NCT06939101
Title: Self-efficacy for Interprofessional Experiential Learning Through an International Service Trip: a Mixed-methods Study
Brief Title: Self-efficacy for Interprofessional Experiential Learning Through an International Service Trip
Status: Completed | Type: Observational
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, William Sit, Clinical Professor, Texas Woman's University
Other Study IDs: IRB-FY2024-248
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: interdisciplinary; Collaboration; education; interaction; evaluation and feedback

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: self-efficacy training — The principal investigator will supervise students and build this program to increase occupational, physical, and speech therapy student participation. There are two one-hour briefing meetings for onboarding to promote self-efficacy preparation and six 1-2 hours of debriefing after each clinical day.

SUMMARY:
This pilot mixed-methods educational study examines the impact of interprofessional experiential learning on self-efficacy during a service trip to Guatemala. Methods: Fourteen participants were recruited from occupational therapy, physical therapy, and speech pathology students at a university. They engaged in a 9-day international interprofessional learning service trip and completed pre- and post-surveys with open-ended questions to measure and reflect on the impact of service trips on self-efficacy.

DETAILED DESCRIPTION:
Description of the service trip The principal investigator is spearheading an education abroad trip to Guatemala involving TWU doctoral entry-level occupational therapy, doctoral physical therapy, and master speech therapy students, building on the program's participation in 2023. The principal investigator will supervise students and build this program to increase occupational, physical, and speech therapy student participation. There are two one-hour briefing meetings for onboarding to promote self-efficacy preparation. The aim is to enhance occupational, physical, and speech therapy student involvement, with the opportunity for subjects to earn credit for Fieldwork I. Organized in collaboration with Hearts in Motion (HIM), an organization dedicated to providing care in areas of need, the 9-day trip from Friday, May 17 to Sunday, May 26, 2024, focuses on improving subjects' self-efficacy for interprofessional experiential learning by offering therapy services to underserved areas in Guatemala. Guatemala is one of the most populated countries in Latin America, and 59.3% of the population lives in poverty. The HIM organizes where the subjects go each day. Upon arrival at a site, the group will break into groups of 2-3 subjects to see each patient, one at a time. Sometimes the subjects are at one of the established therapy clinics HIM runs; sometimes, the subjects have what are called "pop-up" clinics, which is when the subjects go to a town and provide therapy services in a space HIM provides for the subjects (not a clinic; it's usually a church, school, gym, etc.). Every one of the six clinical days has about 30 minutes of briefing before the clinical trip to promote self-efficacy interaction and 60 minutes of debriefing with the PI after the trip for reflection in interprofessional evaluation and feedback on self-efficacy.

Recruitment will begin with the co-investigator sending an email to all TWU students within the occupational, physical, and speech therapy departments regarding the service trip. Following that message, an email from the principal researcher will be sent to the potential subjects who have committed to participating in the trip (see recruiting email attachment in Section 6: subject recruitment), subjects will complete a pre-trip online survey using Qualtrics, assessing their self-efficacy for interprofessional experiential learning. To facilitate post-trip survey matching, subjects will input four digits, comprising their first name initial, two digits of their birthday (01-31), and the last digit of their phone number. All subjects will partake in the same service trip, and upon their return to the United States, they will repeat the survey to evaluate the impact of experiential learning on their confidence levels. Subsequently, subjects will be invited by the PI via a post-trip email to complete an online post-trip survey, compare their self-efficacy for interprofessional experiential learning post-trip, and respond to six open-ended questions about motivation, knowledge, skills, and satisfaction arising from their learning experiences and reflection. Those who have chosen not to participate will receive the email, but they can only accept it if it is applicable.

Throughout the study, communication will be via email, with no video or audio components, allowing subjects to choose a comfortable and private location for survey completion. The estimated time commitment for subjects is 15 minutes for the pre-trip survey and 25 minutes for the post-trip survey, totaling 40 minutes for the entire study. The qualitative method will yield descriptive data from the six open-ended questions only in the post-trip survey created by the PI on subjects' perceived experiences and self-efficacy growth, while closed-ended survey questions will be quantitatively analyzed using SPSS with a repeated measures ANOVA test. The principal investigator and a research team member will analyze qualitative data from open-ended survey questions using a co-coding method with the PI and research team members for rigor and trustworthiness to enhance interrater reliability. A co-principal investigator will be consulted if a disagreement arises between the PI and two research members to come to a consensus during the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old. Plan to attend the service trip in Guatemala. Interprofessional students from the School of Physical Therapy, Occupational Therapy, and Speech Pathology.

Students who have treated clients with other professionals on the service trip.

Exclusion Criteria:

* Students from other academic institutions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The potential subjects in this study consist of approximately 25 Texas Woman's University students from the Occupational Therapy (OT), Physical Therapy (PT), and Speech Therapy (ST) departments.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Self-efficacy intereprofessional experiential scale and six open end questions | pre-post trip surveys about 2 weeks apart
  The pre-trip test consists of five demographic questions. A repeated survey consisting of 16 was developed, tested, and administered pre- and post-trip to measure the dependent variables, which is a highly validated and reliable measurement tool created by Mann. et al. . The confidence variables were measured on a ten-choice Likert scale to reduce central tendency bias. Confidence level was assessed through multiple-choice questions formatted to elicit clinical reasoning based on two factors, including interprofessional interaction and interprofessional evaluation and feedback. The six open-ended questions in the post-trip survey were developed by the research team and reviewed by a biostatistician using survey methods.

CONTACTS AND LOCATIONS:
Overall Officials: william sit, PhD, Principal Investigator — Texas Woman's University (TWU)
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No